CLINICAL TRIAL: NCT07319507
Title: Immediate Remote Effects of Myofascial Release Versus the Fascial Distortion Model on Flexibility and Postural Control Via the Superficial Back Line: A Randomized Pilot Study
Brief Title: Immediate Effects of Calf and Plantar Fascia Manual Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JiYoung Kim (Other)
Responsible Party: Sponsor-Investigator, JiYoung Kim, Adjunct Professor, Physical Therapy, Kyungnam University
Organization: Kyungnam University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JYK-2025-01
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Musculoskeletal Function
Keywords: Myofascial release; Fascial distortion model; Manual therapy; Postural control; Flexibility; Calf muscle and plantar fascia
MeSH Terms: interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel intervention groups, receiving either myofascial release or the fascial distortion model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial Release (Experimental): Participants receive myofascial release to the calf muscles and plantar fascia.
  Interventions: Other: Myofascial Release
- Fascial Distortion Model (Experimental): Participants receive Fascial Distortion Model treatment to the calf muscles and plantar fascia.
  Interventions: Other: Fascial Distortion Model

INTERVENTIONS:
Other: Myofascial Release — Myofascial release applied to the calf muscles and plantar fascia using gentle, sustained manual pressure.
  Arms: Myofascial Release
Other: Fascial Distortion Model — Fascial Distortion Model techniques applied to the calf muscles and plantar fascia using targeted manual pressure.
  Arms: Fascial Distortion Model

SUMMARY:
This study investigated the immediate effects of two manual therapy approaches, myofascial release and the fascial distortion model, applied to the calf and plantar fascia in healthy adults. Participants were randomly assigned to one of the two intervention groups. Flexibility, balance, and postural control were assessed before and after the intervention to examine potential remote effects along the superficial back line. The purpose of this study was to compare the short-term functional effects of these two manual therapy techniques.

DETAILED DESCRIPTION:
This randomized pilot study included healthy adult participants who were assigned to either a myofascial release group or a fascial distortion model group. Manual therapy was applied to the calf muscles and plantar fascia of the dominant lower extremity. Outcome measures related to flexibility, balance, and postural control were assessed immediately before and after the intervention. The study was designed to explore short-term functional changes and to compare the effects of two different manual therapy techniques.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults in their 20s (aged 20-29 years).
* Individuals without current musculoskeletal pain or functional limitations.
* Individuals able to understand the study procedures and provide informed consent.

Exclusion Criteria:

* History of lower extremity injury within the past 6 months.
* Previous experience with plantar fascia manual therapy.
* Presence of balance disorders or neurological impairments.

Ages: 20 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Weight-Bearing Lunge Test (WBLT) | Immediately before and immediately after the intervention
  The Weight-Bearing Lunge Test was used to assess ankle dorsiflexion range of motion by measuring the maximum distance (cm) from the great toe to the wall while maintaining heel contact.

SECONDARY OUTCOMES:
Straight Leg Raise Test (SLR) | Immediately before and immediately after the intervention
  The Straight Leg Raise test was used to assess hamstring flexibility. With the participant in a supine position, the hip was passively flexed with the knee fully extended, and the maximum hip flexion angle (degrees) was measured using a goniometer.
Functional Reach Test (FRT) | Immediately before and immediately after the intervention
  The Functional Reach Test was used to assess dynamic balance. Participants stood upright and reached forward as far as possible without stepping or losing balance. The distance (cm) between the starting position and the maximal forward reach was recorded.
Single-Leg Hop for Distance Test (SLHD) | Immediately before and immediately after the intervention
  Single-Leg Hop for Distance Test (SLHD)
Bunkie Test (BT) | Immediately before and immediately after the intervention
  The Bunkie Test was used to assess lower-extremity and trunk muscular endurance related to the Superficial Back Line. Participants maintained the test position as long as possible, and the holding time (seconds) was recorded.
Finger-to-Floor Distance Test (FFD) | Immediately before and immediately after the intervention
  The Finger-to-Floor Distance test was used to evaluate trunk and posterior chain flexibility. Participants bent forward from a standing position with knees extended, and the vertical distance (cm) between the fingertips and the floor was measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Gyeongsangnam-do, Changwon, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No